CLINICAL TRIAL: NCT03231956
Title: Noninvasive Hemodynamic Monitoring Utilizing ClearSight TM System in Suspected Sepsis Patients Presenting to the Emergency Department (CLEAR SEPSIS)
Brief Title: CLEAR Sepsis Clinical Study
Acronym: CLEAR Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-04
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory specimens to be collected include blood and will be analyzed for lactate at a central clinical research laboratory (WSU Integrative Biosciences, Detroit, MI). Additionally, plasma samples will be obtained for and stored at the WSU Biobank to support potential future clinical and translational research. Samples for the purpose of the WSU Biobank are optional to the clinical research participant and will not adversely affect participation in the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Group 0: Control Sepsis Mimic Group (minor infections or asthma/COPD exacerbations) venous blood lactate levels are not required for this subgroup.
  Interventions: Device: ClearSight™ / EV1000NI Clinical Platform
- Group 1: Suspected infection plus Initial Venous Blood Lactate ≥ 0 - 1.9 mmol/dL
  Interventions: Device: ClearSight™ / EV1000NI Clinical Platform
- Group 2: Suspected infection plus Initial Venous Blood Lactate ≥ 2.0 - 3.9 mmol/dL
  Interventions: Device: ClearSight™ / EV1000NI Clinical Platform
- Group 3: Suspected infection plus Initial Venous Blood Lactate ≥ 4.0 mmol/dL
  Interventions: Device: ClearSight™ / EV1000NI Clinical Platform

INTERVENTIONS:
Device: ClearSight™ / EV1000NI Clinical Platform — Noninvasive Hemodynamic Monitoring utilizing ClearSight TM System

SUMMARY:
To investigate the relationship between initial ClearSight™ derived hemodynamic parameters and outcomes (death, ongoing organ dysfunction or delayed ICU admission) in patients with acute infection and possible sepsis, with a focus on venous blood lactate (< 2.0, 2.0-3.9, and ≥ 4.0 mmol/dL) and hemodynamic subgroups, using ED patients presenting with minor infections or asthma/COPD exacerbations as controls (henceforth referred to as Sepsis Mimic Group).

ELIGIBILITY:
Venous Blood Lactate Groups

Inclusion Criteria:

* ≥ 18 years of age at the time of enrollment
* Any combination of acute symptoms and signs that the treating ED physician, after initial history and physical examination, attributes to a systemic infection
* ED Physician confirms likely hospital admission (> 50%) due to suspicion of infection
* ED Physician confirms intention to order both blood cultures and venous blood lactate levels
* Ability to enroll patient and begin ClearSight™ monitoring within three (3) hours of ED presentation

Exclusion Criteria:

* Initial venous blood lactate measured > 3 hours after ED arrival
* Pre-existing infection for which patient is being treated with antibiotics as an outpatient
* Prisoners
* Pregnant women
* Any previous medical condition with life expectancy of < 3 months (patients with ESRD and heart failure are not excluded)
* DNR or comfort care order preexisting to ED visit or established in the ED
* Palliative care or hospice consult in the ED
* Known severe aortic insufficiency
* Known history of Raynaud's disease
* Poor follow-up candidate in the opinion of the Investigator
* Current or planned enrollment in an investigational trial that in the opinion of the Investigator may significantly affect hemodynamic data collection.

Control Sepsis Mimic

Inclusion Criteria:

* ≥18 years of age at the time of enrollment
* Presents to the ED with a chief complaint consistent with a minor infection (upper respiratory infection, soft tissue infection, viral infection) or an asthma or COPD exacerbation on whom the treating physician is not ordering labs for blood cultures or lactate levels
* Ability to enroll patient and begin ClearSight™ monitoring within three (3) hours of ED presentation.

Exclusion Criteria:

* Pre-existing infection for which patient is being treated with antibiotics as an outpatient
* Prisoners
* Pregnant women
* Any previous medical condition with life expectancy of < 3 months (patients with ESRD and heart failure are not excluded)
* DNR or comfort care order preexisting to ED visit or established in the ED
* Palliative care or hospice consult in the ED
* Known severe aortic insufficiency
* Known history of Raynaud's disease
* Poor follow-up candidate in the opinion of the Investigator
* Current or planned enrollment in an investigational trial that in the opinion of the Investigator may significantly affect hemodynamic data collection.
* Treating physician is planning on ordering either a lactate or blood cultures on the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute infection and possible sepsis, with a focus on venous blood lactate (< 2.0, 2.0-3.9, and ≥ 4.0 mmol/dL) and hemodynamic subgroups, using ED patients presenting with minor infections or asthma/COPD exacerbations as controls (henceforth referred to as Sepsis Mimic Group).
Sampling Method: Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | Within 72 hours of presentation
  Increase in modified Sequential Organ Failure Assessment (mSOFA) score ≥ 1 resulting in ICU admission / death.
Venous Blood Lactate clearance | Within 24 and 72 hours of presentation
  Venous Blood Lactate clearance
Length of Stay | 30 days
  Emergency Department length of stay, ICU length of stay, and Hospital length of stay
Recidivism | 30 days
  Recidivism within 30 days of the index hospital visit

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Beaumont Hospital, Troy, Troy, Michigan

IPD SHARING:
Plan to Share IPD: No